CLINICAL TRIAL: NCT06715800
Title: Symptomatic Relief of Sore Throat With Functional Honey: A Randomized Controlled Trial
Brief Title: Honey Against Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ali Timucin ATAYOGLU, Assoc. Prof., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.29934
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Sore Throat; Honey
Keywords: Sore throat; Apitherapy; Functional Honey
MeSH Terms: conditions — Pharyngitis | interventions — Honey; High Fructose Corn Syrup

STUDY DESIGN:
Intervention Model Description: Double blind, Randomized, Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- H1 Thyme honey group (Active Comparator): The group who applied with the complaint of sore throat was cultured and given thyme honey in addition to drug treatment.
  Interventions: Dietary Supplement: Honey
- H2 Yuksekova honey group (Active Comparator): The group who applied with the complaint of sore throat was cultured and given Yuksekova honey in addition to drug treatment.
  Interventions: Dietary Supplement: Honey
- H3 Chestnut honey group (Active Comparator): The group who applied with the complaint of sore throat was cultured and given chestnut honey in addition to drug treatment..
  Interventions: Dietary Supplement: Honey
- H4 Linden honey group (Active Comparator): The group who applied with the complaint of sore throat was cultured and given linden honey in addition to drug treatment.
  Interventions: Dietary Supplement: Honey
- H5 Pine honey group (Active Comparator): The group who applied with the complaint of sore throat was cultured and given pine honey in addition to drug treatment.
  Interventions: Dietary Supplement: Honey
- H6 Plasebo group (Placebo Comparator): The group who applied with the complaint of sore throat was cultured and given plasebo in addition to drug treatment.
  Interventions: Dietary Supplement: Honey

INTERVENTIONS:
Dietary Supplement: Honey — Functional content analyses were performed to identify the specific properties of the different types of honey used.
  Other Names: Thyme Honey; Southeastern Anatolia; Chestnut honey; Linden honey; Pine honey; sugar syrup

SUMMARY:
Objective: The aim of this study is to investigate the symptomatic efficacy of oral use of different functional honeys in patients complaining of sore throat.

Materials and Methods: In the preclinical phase of the study, a total of 1000 samples of honey were examined, and the honeys were subjected to physicochemical and microbiological analyses. Based on their functional properties, five different groups of honey were determined. These are thyme honey with high antioxidant capacity, Yüksekova with high antimicrobial activity, chestnut honey with high organic acid amount, linden honey with high enzymatic and pine honey with high anti-microbial, antioxidant and phenolic compounds and enzymes. In the clinical phase of the study, patients receiving conventional treatment were randomly assigned to receive either one of five different types of honey or a honey-like food product in addition to their treatment. They were instructed to use 15 grams twice daily for 10 days. Patients were assessed on the 1st, 3rd, 7th, and 10th days for symptoms and complaints such as sore throat, difficulty swallowing, sensation of throat swelling, weakness, and fatigue.

ELIGIBILITY:
Inclusion Criteria: Adults presenting with sore throat symptoms due to an upper respiratory infection (URI) within the last four days were included in the study. A total of 300 patients over 18 years of age, who were prescribed necessary medication and exhibited signs and symptoms of sore throat, were enrolled.

Exclusion Criteria: Exclusion criteria included a history of diabetes, pollen or bee allergies, and aversion to honey. Participants were required not to use any additional products outside of those provided by the researchers during the study period. Written informed consent was obtained from all participants, who were then randomly assigned to either the study or control group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Clinical Symptome | 10 days
  Symptom Evaluation: On days 3, 7, and 10, patients were assessed for throat pain, difficulty swallowing, throat swelling, and fatigue/malaise.
  Throat Pain: Assessed using a Numeric Rating Scale (NRS) (0: no pain, 10: very painful).
  Difficulty Swallowing: Assessed using a NRS (0: no difficulty, 10: very difficult).
  Throat Swelling Sensation: Assessed using a NRS (0: no swelling, 10: severe swelling sensation).
  Fatigue/Malaise: Assessed using a NRS (0: no fatigue, 10: severe fatigue).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided